CLINICAL TRIAL: NCT02225236
Title: Improving Self-regulation & School Readiness in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Brady Education Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FP00006613
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Executive Dysfunction
Keywords: executive functioning; metacognition; self-regulation; preschoolers
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classroom Intervention (Experimental): The intervention focuses on training executive functioning (e.g., working memory and inhibition) and metacognition (i.e., the ability to predict, check, monitor, coordinate and control cognitive operations) using play activities and structured language and reinforcement.
  Interventions: Behavioral: Classroom Intervention
- No treatment control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Classroom Intervention
  Arms: Classroom Intervention

SUMMARY:
This project will develop and evaluate the initial effectiveness of an intervention training executive functioning, metacognition, and self-regulation in preschoolers attending certain high poverty Cincinnati preschools. Studies show that these skills are critical for school performance, and that children with better executive functioning have better long term outcomes. It is also important to intervene early when children are most likely to profit because their brains are rapidly developing. There are some promising programs targeting these skills in preschoolers, but few are available to teachers for implementation in the classroom setting. The specific aims of this study are: 1) to adapt a promising clinic-based program for the preschool classroom environment, and 2) to test the feasibility and initial impact of the adapted program on executive functioning and school readiness in schools with a high proportion of children from low income families.

DETAILED DESCRIPTION:
We propose to translate a promising intervention, Executive-function Training for Attention and Metacognition (ETAM), originally developed for use in a clinic setting, to be delivered in the school setting, ultimately by teachers. Specifically, we propose to develop a curriculum that can be added to the classroom curriculum which will target the development of self-regulation and metacognition in preschoolers. Thus the purpose of the study is to 1) develop a teacher training program based on the principles we have found to be effective in a parent-based intervention and 2) test the feasibility and initial efficacy (i.e., reduced disruptive behaviors and increased school readiness) of the program in children from low income families. We will randomly assign 6 preschools to receive the teacher training component and 6 schools to serve as a control group (i.e., will not receive the intervention). We will conduct assessments on all preschoolers in the classroom prior to delivering the teacher training (i.e., beginning of the school year), provide the training to preschoolers in classrooms randomized to the active intervention group, and then conduct assessments at the end of the school year. Our primary aims are to assess the feasibility of a program designed to train teachers to incorporate the principles of the training program into the daily classroom environment, and to assess whether the program improves executive functioning and functional outcomes [i.e., Attention/Deficit-Hyperactivity Disorder (ADHD) symptoms, academic readiness, social competence], as compared to outcomes of children in the control schools. Although study personnel will be responsible for delivery of the intervention, preschool teachers will be closely involved in the process to provide ongoing feedback regarding the study intervention.

ELIGIBILITY:
Inclusion Criteria:

All children in preschool classrooms in selected schools.

Exclusion Criteria:

None

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function-Preschool Version | Outcome assessment (~9 months after initial assessment)
  Parents and teachers will complete this rating scale assessing executive function behaviors in the home and school environments, yielding T-scores on several subscales, including Inhibit, Shift, Emotional Control, Working Memory, Plan/Organize, Inhibitory Self-Control Index, Flexibility Index, Emergent Metacognition Index, and a Global Executive Composite. The scale has adequate reliability and validity as assessed in two- to five-year-olds

SECONDARY OUTCOMES:
Clinical Evaluation of Language Fundamentals - Preschool, Second Edition - Concepts and Following Directions | Outcome evaluation (~9 months after baseline evaluation)
  The Concepts and Following Directions subtest is a measure of auditory and visual attention. This subtest requires the child to interpret, recall, and execute oral commands of increasing length and complexity that contain concepts of functional language. A subscale score is computed for Concepts and Following Directions. Across ages (i.e., 3- to 7-year-olds), internal consistency ranged from .78 to .85 with an average of .82.
NEPSY- Attention/Executive Function subtests | Outcome (~9 months after baseline evaluation)
  The Visual Attention subtest is a measure of inhibition, scanning, vigilance, and impulsivity. This subtest is divided into two tasks (e.g., cats and faces, or bunnies and cats). The child is shown an exemplar at the top of the page (e.g., bunny) and is asked to circle all the bunnies amongst a number of other stimuli on the rest of the page as quickly as possible. The Statue subtest is a measure of motor persistence and inhibition. The child is asked to assume a pose and remain in it with their eyes closed for 75 seconds, ignoring distractors occurring at regular intervals. A subscale score is computed for each subtest. Reliabilities for the NEPSY at ages 3 through 7 are > .70.
Shape School | Outcome (~9 months after baseline evaluation)
  This assessment is a developmentally appropriate task developed for preschoolers assessing inhibition and switching. The child is presented with a colorful storybook of colorful circle and square figures and is administered 4 conditions (control, inhibit, switch, concurrent/both). In the control condition, the child names the colors of the figures as fast as possible. In the inhibit (response suppression) condition, the child only named the colors of the figures with happy faces and not frustrated faces. In the switch (attention control) condition, the child names the shapes of figures wearing hats. In the concurrent condition, the child is asked to name the figures (color or shape), who were both wearing hats and had happy faces. Cronbach's alpha coefficients for each condition exceeds 0.71.
Swanson, Kotkin, Agler, M-Flynn, Pelham (SKAMP) Teacher Rating Scale | Outcome (~9 months after baseline evaluation)
  Teachers will be asked to complete the SKAMP to measure impairments in classroom functioning related to disruptive behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Tamm, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Schools in the Archdiocese of Cincinnati to be determined, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Tamm L, Peugh J. Concordance of teacher-rated and performance-based measures of executive functioning in preschoolers. Child Neuropsychol. 2019 Apr;25(3):410-424. doi: 10.1080/09297049.2018.1484085. Epub 2018 Jun 14. PMID 29902951